CLINICAL TRIAL: NCT03672552
Title: Implementing the Frazier Free Water Protocol to Improve Hydration and Quality of Life in Long Term Care Residents
Brief Title: Using Plain Water With Oral Care to Increase Hydration for Long Term Care Residents With Disordered Swallowing
Acronym: FFWP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: Eastern Health (Other); Newfoundland and Labrador Support for Patient-Oriented Research (Unknown)
Responsible Party: Principal Investigator, Roberta DiDonato, Adjunct Professor, Faculty of Science and Medicine, Research Director Anesthesiology, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018.162
Record Dates: First submitted 2018-09-08; First posted 2018-09-14 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Dysphagia; Respiratory Tract Infections
Keywords: Aspiration pneumonia; Dementia; Dysphagia; Oral hygiene; Long-term care; Frazier Free Water
MeSH Terms: conditions — Deglutition Disorders; Respiratory Tract Infections; Pneumonia, Aspiration; Dementia

STUDY DESIGN:
Intervention Model Description: All study participants will have assessments for swallowing and oral hygiene. The intervention group will have a dental hygiene cleaning and supervised tooth brushing before taking plain, thin (unmodified) water and between meals. The control group will continue with standard oral care and the agreed upon diet texture and fluid modifications.
Who Masked: Participant
Masking Description: Participants may identify with the study receiving more oral care than previously but not know if they are in the intervention or control group. Clinicians performing swallowing and oral health assessments will not know which participants are randomly assigned to groups. Nursing staff will be performing daily care on all participants as specified in daily nursing protocols and may have more oral care but may not identify whether a participant is in the intervention or control group except some staff will be adding supervised brushing before plain (thin) water and between mealtimes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FFWP and Improved Oral Care (Experimental): Receiving dental hygienist cleaning with supervised tooth brushing and FFWP (plain, unmodified water).
  Interventions: Other: FFWP and Improved Oral Care
- Standard Care (No Intervention): This group has assessments and standard oral care with no dental hygienist cleaning, no FFWP or supervised tooth brushing and continuing with agreed upon diet texture and fluid modification.

INTERVENTIONS:
Other: FFWP and Improved Oral Care — The FFWP with dental hygiene participants will have assessments for swallowing and oral health then proceed to have a dental hygienist cleaning. This intervention group will have supervised and assisted tooth brushing by nursing staff before taking plain (thin) unmodified water and between meals.
  Other Names: Dental hygienist intervention and supervised tooth brushing
  Arms: FFWP and Improved Oral Care

SUMMARY:
The Frazier Free Water Protocol (FFWP) using plain, thin (unmodified) water is an accepted method to increase fluid intake and hydration in older adults with disordered swallowing and dementia.This study aims to take an interdisciplinary approach to see if the FFWP with improved oral care can be introduced in a long term care (LTC) setting comparing an intervention group with a control group receiving standard oral care, to prevent respiratory infections.

DETAILED DESCRIPTION:
The investigators will recruit a convenience sample of 36 participants from a single long-term care facility. Participants will be randomly assigned into control or intervention groups. Both groups will be assessed at study onset for swallowing and oral health and continue with agreed upon diet texture and fluid modifications. The intervention group (FFWP and improved oral hygiene) will receive a dental hygienist cleaning at onset of the study and have supervised tooth brushing before thin water between meals. The control group will continue with standard oral care and offered the full dental hygienist cleaning at the end of the study. If findings indicate no difference between groups on outcome measures (eg. respiratory illness, hydration, nutrition) then the intervention is considered efficacious in long-term care residents. If improvements in outcome measures are evident for the treatment relative to the control group, then this intervention may provide opportunity for improved healthcare and cost-savings.

ELIGIBILITY:
Inclusion Criteria:

* Long Term Care Residents with moderate to severe swallowing difficulty and modified texture diet; or have a dry mouth and thirsty most of the time by report of patient participant, family or staff.

Exclusion Criteria:

* Participant Resident taking part in another study; participant finished another study in last 30 days prior to this study; Participant has dental pain or waiting to see a dentist for pain and discomfort; Participant has current chest infection including pneumonia or is prone to chest infections with more than one episode per year; Participant is unable to tolerate assessments and oral care.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Chest Infections | Change from baseline (Day-0 to 90 days)
  To determine whether the Frazier Free Water Protocol (FFWP) with improved oral care will decrease risk of respiratory illness events (eg. chest congestion, fever, etc.) for long term care residents by numbers of documented cases of upper and lower respiratory illnesses and hospital admissions over a 90-day duration.

SECONDARY OUTCOMES:
Incidence of positive experience with FFWP intervention. | Change from baseline (Day 0-90 days)
  Analysis of participant experience with FFWP intervention over the 90-day study period by scaled responses to feedback question: Did you feel this was a positive experience? Responses range from Strongly Agree, Agree, Disagree, Strongly Disagree and Neither Agree or Disagree.
Change in Hydration | Change from baseline (Day-0 to 90 days)
  To assess change in hydration associated with FFWP intervention measured by lab values for electrolytes, BUN (Blood, Urea, Nitrogen) and Creatinine obtained over the 90-day study period.
Change in Nutrition. | Change from baseline (Day 0 to 180 days)
  To assess change in nutrition associated with FFWP intervention measured by lab values for albumin, BUN (Blood, Urea, Nitrogen) and Creatinine obtained over the 90-day study period.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta M DiDonato, PhD, Principal Investigator — Memorial University of Newfoundland
Locations (1):
- Eastern Health-Pleasant View Towers, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No
Data sharing guarded by privacy legislation and will require special application. Some documentation or research materials without participant data or identification may be shared.

REFERENCES:
- [Result] Gillman A, Winkler R, Taylor NF. Implementing the Free Water Protocol does not Result in Aspiration Pneumonia in Carefully Selected Patients with Dysphagia: A Systematic Review. Dysphagia. 2017 Jun;32(3):345-361. doi: 10.1007/s00455-016-9761-3. Epub 2016 Nov 23. PMID 27878598
- [Result] Azarpazhooh A, Leake JL. Systematic review of the association between respiratory diseases and oral health. J Periodontol. 2006 Sep;77(9):1465-82. doi: 10.1902/jop.2006.060010. PMID 16945022
- [Result] Cabre M, Serra-Prat M, Palomera E, Almirall J, Pallares R, Clave P. Prevalence and prognostic implications of dysphagia in elderly patients with pneumonia. Age Ageing. 2010 Jan;39(1):39-45. doi: 10.1093/ageing/afp100. Epub 2009 Jun 26. PMID 19561160
- [Result] Forsell M, Kullberg E, Hoogstraate J, Johansson O, Sjogren P. An evidence-based oral hygiene education program for nursing staff. Nurse Educ Pract. 2011 Jul;11(4):256-9. doi: 10.1016/j.nepr.2010.11.017. Epub 2010 Dec 23. PMID 21185232
- [Result] Wirth R, Dziewas R, Beck AM, Clave P, Hamdy S, Heppner HJ, Langmore S, Leischker AH, Martino R, Pluschinski P, Rosler A, Shaker R, Warnecke T, Sieber CC, Volkert D. Oropharyngeal dysphagia in older persons - from pathophysiology to adequate intervention: a review and summary of an international expert meeting. Clin Interv Aging. 2016 Feb 23;11:189-208. doi: 10.2147/CIA.S97481. eCollection 2016. PMID 26966356
- [Result] Agarwal E, Marshall S, Miller M, Isenring E. Optimising nutrition in residential aged care: A narrative review. Maturitas. 2016 Oct;92:70-78. doi: 10.1016/j.maturitas.2016.06.013. Epub 2016 Jun 23. PMID 27621242
- See also: The Prevalence of Dysphagia in Long-Term Care Facility [Thesis]; Memorial University, St. John's , NL — http://research.library.mun.ca/id/eprint/11694